CLINICAL TRIAL: NCT06927076
Title: Investigating the Role of the Psychedelic Experience in the Antidepressant Response in Patients With Major Depression: a Placebo-controlled Factorial Trial With DMT Masked With Propofol (DMT4D-Study)
Brief Title: Antidepressant Response of DMT Masked With Propofol
Acronym: DMT4D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-02312;am24Liechti6
Record Dates: First submitted 2025-04-04; First posted 2025-04-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder; Psychedelic Experiences
Keywords: N,N-dimethyltryptamine (DMT); neuroplasticity
MeSH Terms: conditions — Depressive Disorder, Major | interventions — N,N-Dimethyltryptamine; Propofol

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind (DMT vs placebo), placebo-controlled, 2x2 factorial parallel group design. Participants are randomly assigned to DMT or placebo (double-blinded) under either sedation with propofol or no sedation (sinlge-blinded).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: DMT and placebo will be administered in a double-blind fashion. However, investigators immediately involved in the treatment of the specific patient will be informed whether the assignment involves propofol or not. Participants will not be informed about the propofol assignment (single-blind).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DMT without sedation (Experimental): DMT without sedation (propofol)
  Interventions: Drug: N,N-Dimethyltryptamine; Procedure: no sedation
- DMT with sedation (Experimental): DMT with sedation (propofol)
  Interventions: Drug: N,N-Dimethyltryptamine; Procedure: Propofol
- Placebo without sedation (Placebo Comparator): Placebo (double-blind) without sedation (propofol)
  Interventions: Drug: Placebo; Procedure: no sedation
- Placebo with sedation (Placebo Comparator): Placebo (double-blind) with sedation (propofol)
  Interventions: Drug: Placebo; Procedure: Propofol

INTERVENTIONS:
Drug: N,N-Dimethyltryptamine — administration of a 2mg/min DMT perfusion over 20 min
  Other Names: DMT
  Arms: DMT with sedation; DMT without sedation
Drug: Placebo — administration of a placebo perfusion over 20 min
  Arms: Placebo with sedation; Placebo without sedation
Procedure: Propofol — 30 min propofol sedation
  Arms: DMT with sedation; Placebo with sedation
Procedure: no sedation — no sedation
  Arms: DMT without sedation; Placebo without sedation

SUMMARY:
The aim of this study is to elucidate if the anti-depressive effect of N,N-dimethyltryptamine (DMT) is based on a biological mechanisms including neuroplasticity and anti-inflammatory effect or due to the subjective psychedelic experience.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) affects nearly 20% of people, but current treatments-both pharmacological and psychotherapeutic-have limited efficacy, especially for mild to severe cases. Psychedelics like LSD, psilocybin, and DMT are being explored as alternative therapies, with studies showing promising antidepressant effects. However, it is unclear whether these benefits stem from their acute subjective (psychedelic) experience or from biological mechanisms like neuroplasticity and anti-inflammatory effects.

This study aims to determine if the antidepressant effects of DMT occur independently of its psychedelic experience. To test this, DMT will be administered under sedation (with propofol) to mask subjective effects, as well as without sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must meet DSM-5 criteria for MDD of at least moderate severity (MADRS>20).
2. Participants either currently do not use antidepressants or are treated with a stable dose for at least 4 weeks prior to randomization.
3. Age ≥ 21 years old.
4. Sufficient understanding of the German language.
5. Able to understand the study procedures and risks and willing to adhere to the protocol and sign the consent form.
6. Willing not to drive or operate heavy machinery on the treatment day.
7. Willing to refrain from more than 7 standard alcoholic drinks a week, more than 10 cigarettes a day, more than 2 cups of coffee a day, and any illicit substances during study participation.
8. Willing to use effective contraceptive measures throughout study participation.

Exclusion Criteria:

1. Past or present bipolar or psychotic disorder, including depressive disorder with psychotic features.
2. First-degree relative with a psychotic or bipolar disorder.
3. Significant prodromal psychotic symptoms (Prodromal Questionnaire-16 symptoms ≥ 6).
4. Psychiatric condition judged to be incompatible with establishment of rapport with study team members and/or safe exposure to DMT, e.g. diagnosed or suspected borderline personality disorder.
5. Current post-traumatic stress disorder or acute stress reaction due to a traumatic event.
6. Post-partum depression.
7. Pregnant or breastfeeding women.
8. Current or recent history of significant suicide ideation or suicide behavior within the past 6 months.
9. Current severe substance use disorder other than nicotine.
10. Planned ketamine, other psychedelic, or electroconvulsive treatment or any such treatment within the past 3 months.
11. Any lifetime use of DMT, use of any other psychedelics within last 3 month or lifetime use of any other psychedelics more than 15 times.
12. Patients who are treated with neuroleptics or known antagonists of 5-HT2 receptors or monoamine oxidase inhibitors (MAOI) and are not able/willing to pause.
13. Increased risk for adverse reactions to propofol or soja products.
14. Increased risk for aspiration.
15. Increased risk for difficult mask ventilation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
long term changes in depressive symptoms (MADRS) | baseline (before intervention) and on day 14 post-intervention
  Changes in depressive symptoms will be assessed using Montgomery-Asberg-Depression Rating Scale (MADRS). The MADRS is a ten-item questionnaire widely used to measure severity of depressive symptoms during the last week. Total score (range 0-60); higher scores indicate greater depression severity.

SECONDARY OUTCOMES:
Short term changes in depressive symptoms (MADRS) | Baseline (before intervention) and on day 1, 3 and 7 post-intervention
  Changes in depressive symptoms will be assessed using Montgomery-Asberg-Depression Rating Scale (MADRS). The MADRS is a ten-item questionnaire widely used to measure severity of depressive symptoms during the last week. Total score (range 0-60); higher scores indicate greater depression severity.
Changes in depressive symptoms (BDI) | Baseline (before intervention) and on day 1, 3, 7 and 14 post-intervention
  Changes in depressive symptoms will be assessed using Beck Depression Inventory (BDI) questionnaire. Total score (range 0-63); higher scores indicate more severe depressive symptoms.
Changes in anxiety (STAI) | Baseline (before intervention) and on day 1, 3, 7 and 14 post-intervention
  Changes in anxiety will be assessed using the self-reported State-Trait Anxiety Inventory (STAI) questionnaire. Separate total scores for State Anxiety (S-Anxiety) and Trait Anxiety (T-Anxiety) (each range 20-80); higher scores indicate greater anxiety.
Changes of clinical global impression (CGI-S) | Baseline (before intervention) and on day 1, 3, 7 and 14 post-intervention
  The clinical global impression (CGI) is an instrument for the assessment of the patient's overall functioning both before and after starting the treatment.
  Severity of Illness (CGI-S): Rated on a 7-point scale (1 = normal, 7 = among the most extremely ill).
Changes of clinical global impression (CGI-I) | Baseline (before intervention) and on day 1, 3, 7 and 14 post-intervention
  The clinical global impression (CGI) is an instrument for the assessment of the patient's overall functioning both before and after starting the treatment.
  Improvement (CGI-I): Rated on a 7-point scale (1 = very much improved, 7 = very much worse).
Changes in quality of life (WHOQOL-bref) | Baseline (before intervention) and on day 1, 3, 7 and 14 post-intervention
  Changes in quality of life will be assessed by World Health Organization Quality of life scale (WHOQOL-bref). The WHOQOL-bref is one of the most commonly used self-rating instruments for the assessment of the quality of life and covers different domains of quality of life (physical, psychological, level of independence, social relationships, and environment, and spirituality). Domain scores (Physical, Psychological, Social, Environmental), scaled from 0 to 100; higher scores indicate better quality of life.
Persisting positive and negative effects (PEQ) | On day 14 post-intervention
  Psychedelics have been shown to produce persisting effects on well-being and appreciation of social relationships on the PEQ.This questionnaire will be used at the EOS visit to assess similar persisting effects of the DMT experience in addition to any effects on depressive symptomatology. Subscale scores (e.g., positive attitudes, mood changes, spirituality), typically rated 0-5 or 0-6; higher scores indicate stronger persisting effects.
Acute subjective effects (5D-ASC) | On day 0 post-intervention
  The 5 Dimensions of Altered States of Consciousness (5D-ASC) Scale is a questionnaire containing visual analog scales for 94 items. The instrument contains five scales assessing mood, anxiety, derealization, depersonalization, changes in perception, auditory alterations, and reduced vigilance. Each item of the scale is scored on a 0-100 mm VAS. Scores for 5 dimensions (e.g., Oceanic Boundlessness, Anxious Ego Dissolution), range typically 0-100%; higher scores indicate more intense altered states.
Subjective Effects Rating (SES) | On day 0 pre- and post-intervention
  Participants will be asked by the investigator to repeatedly rate their subjective effects verbally on a Likert scale from 0 to 10 for: "any drug effect", "good drug effect", "bad drug effect", and "fear". Ratings will be performed before and repeatedly after substance administration and will take approximately 30 sec to complete. The time course and maximal ratings (Emax, 0-10) are defined for each rating and Emax values compared between treatments using analysis of variance (ANOVAs). Total and subscale scores (range and subscales vary by implementation); higher scores indicate more intense subjective effects.
Psychedelic Experience Scale (PES) | On day 0 post-intervention
  In the PES, 100-items are rated on a six-point scale. The PES represents a revalidation of the original 100-item States of Consciousness Questionnaire (SOCQ)
Emotional breakthrough inventory (EBI) | On day 0 post-intervention
  The Emotional breakthrough inventory (EBI) is a validated instrument with 6 items to assess the degree of emotional breakthrough as a distinct component of the acute psychedelic experience. Total score (range varies); higher scores indicate stronger emotional breakthrough experiences.
Acute adverse effects | On day 0 post-intervention
  Acute adverse effects wil be assessed by the List of complaints (LC). LC is a self-reporting tool to assess physical and general discomfort. A revised version is used which consists of a 40-item list covering a wide variety of symptoms and complaints that are answered with a four-point intensity-scoring ranging from "not at all" to "strong". Total number or severity of reported somatic and psychological complaints will be evaluated.
Safety events | From day 0 to day 14 post-intervention
  Adverse events will be assessed over the whole study period.
Neuroplasticity | Baseline (before intervention) and on day 14 post-intervention
  brain-derived neurotrophic factor (BDNF), a biomarker for neurogenesis will be quantified in blood samples collected before and 14 days after intervention
Inflammation | Baseline (before intervention) and on day 14 post-intervention
  Interleukin-1 beta (IL-1β) an immunological factor linked to depression will be quantified in blood samples collected before and 14 days after intervention
DMT plasma concentration | On day 0 shortly before the end of the perfusion
  Plasma levels of DMT will be measured once shortly before the end of the perfusion
Expectancy (CEQ) | At Baseline before intervention
  Expectancy will be assessed before the first drug administration. Thus, patients will know at this timepoint whether they get the treatment with or without propofol. To measure expectancy, a modified 2-item version of the Credibility / Expectancy Questionnaire (CEQ) is used. Credibility score (range 3-27).
Expectancy | At Baseline before intervention
  The Stanford Expectations of Treatment Scale (SETS) will evaluate positive and negative expectancies. Expectancy score (range 3-27 or expressed as a probability %).
Mood | At day 0 directly before administration of the study drug
  The Adjective Mood Rating Scale (AMRS) is a self-rating scale assessing current mood states. The AMRS will be used to assess mood before the DMT experience. Positive mood and greater acute well-being is expected to positively enhance the acute DMT effects as similarly shown for other psychedelics. Scores for multiple mood dimensions (e.g., energy, mood, agitation); higher scores reflect greater expression of that dimension.
Personality (NEO-FFI) | At Baseline before intervention
  Personality traits are known to affect subjective responses to psychoactive substances. The NEO Five Factor Inventory (NEO-FFI) will be used during screening to self-assess personality traits. Scores for five domains (Neuroticism, Extraversion, Openness, Agreeableness, Conscientiousness); raw or standardized T-scores.
Personality (TAS) | At Baseline before intervention
  Personality traits are known to affect subjective responses to psychoactive substances. The Tellegen Absorption Scale (TAS) will be used during screening to self-assess personality traits. Total score (range 0-34 or 0-136, depending on version); higher scores indicate greater trait absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Liechti, Prof. Dr. med., Study Director — University Hospital, Basel, Switzerland; Felix Müller, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland